CLINICAL TRIAL: NCT06158997
Title: Safety and Effectiveness of EyePeace on Signs and Symptoms of Dry Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEDEP2023
Record Dates: First submitted 2023-02-06; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Evaporative Dry Eye
Keywords: Dry eye; Eye massage; Diquafosol; Eyepeace
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective, comparative pilot study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masked examiner for all clinical assessments will not involved in the data collection or group allocation procedure for this research. The investigator will not be aware of the two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EyePeace+Heated eye mask group (Experimental): Participants will received the HEM therapy for 10 minutes according to the manufacturer's instructions. This was followed immediately by 10 gentle squeezes of the eyelid massage device on one eye
  Interventions: Device: EyePeace; Device: Heated Eye Mask
- Heated Eye Mask group (Active Comparator): Participants in Heated Eye Mask group will use heated eye mask once.
  Interventions: Device: Heated Eye Mask

INTERVENTIONS:
Device: EyePeace — EyePeace a commercially available for enhancing meibum expression. The flexible, handheld device is made of silicone and provides regulated vertical pressure on closed eyelids (https://www.eyepeace.de). EyePeace will be used to assess its usefulness in improving evaporative dry eye signs and symptoms.
  Other Names: Eye massager
  Arms: EyePeace+Heated eye mask group
Device: Heated Eye Mask — Heated Eye Mask will be used once a day to assess its usefulness in improving evaporative dry eye signs and symptoms.
  Other Names: HEM

SUMMARY:
In this study, the EyePeace an eye massager will be compared with a standard-of-care warm compress treatment with evaporative dry eye disease. The objective is to asses the safety and effectiveness EyePeace eye massager is in relieving the signs and symptoms of evaporative dry eye disease.

DETAILED DESCRIPTION:
A prospective, contralateral-eye trial study compared the effects of Eyepeace+Heated eye mask versus Heated eye mask with dry eye patients. Following 10 min of heated eye mask on both eyes, eyelid massage therapy was applied to the right eye by device. The efficiency was evaluated at baseline (0 mins), 5 minutes (5 mins), 15 minutes (15 mins), and 30 minutes (30 mins) by having the patient perform the eyelid expression massage under the supervision of an ophthalmologist. Non-invasive breakup time (NITBUT), tear meniscus height (TMH), tear-film lipid layer (TFLL), ocular surface temperature (OST), meibomian gland quality (MGQ), meibomian gland expressibility (MGEx), best corrected visual acuity (BCVA), intraocular pressure (IOP), endothelial cell count (ECC), flat-axis keratometry value (K1), steep-axis keratometry value (K2), and central corneal thickness (CCT) were examined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able and willing to comply with the treatment/follow-up schedule
* Bilateral signs and symptoms of dry eye disease or MGD

Exclusion Criteria:

* Treat dry eye with medication or massage or fumigation within 1 month
* The eyelids or intraocular tumor unfavorable pressure
* Previous ocular surgery or trauma
* Barriers to the subjects in the research of ocular surface active allergies, infection or inflammatory bowel disease
* Intraocular pressure is less than 10 mmHg or more than 21 mmHg
* Diabetes or other eye table, healthy body, skin diseases, or diseases of the nervous system;
* Use any may interfere with tears within three months of systemic anti-inflammatory drugs or medicines, such as resistance to anxiety, depression and antihistamines
* The local administration of ophthalmology recent history (in the past 30 days) including antibiotics, steroids and non-steroidal anti-inflammatory drug, or long-term use of local ophthalmic drug
* Researchers determine patients not suitable for this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-03 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Non-invasive tear break-up time | Baseline, 5 min, 15 min, 30 min
  Changes in non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer.
  Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.
Tear Film Lipid Layer | Baseline, 30 min
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan).
Expressibility of meibum grade | Baseline, 5 min, 15 min, 30 min
  Meibum expressibility will be assessed under a slit-lamp:
  Eight meibomian glands in the middle part will be evaluated on a scale of 0 to 3 (0 denoted that all glands expressible; 1 denoted that 3 to 4 glands expressible; 2 denoted those 1 to 2 glands expressible; and 3 denoted that no glands were expressible). The overall score was computed using the mean scores of these eight glands.
Quality of meibum grade | Baseline, 5 min, 15 min, 30 min
  Meibum quality will be assessed under a slit-lamp:
  Five meibomian gland in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste like consistency meibum).

SECONDARY OUTCOMES:
Conjunctival hyperemia (RS score) | Baseline, 5 min, 15 min, 30 min
  Conjunctival hyperemia (RS score) will be assessed by keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 to 4.0.
Conjunctivocorneal epithelial staining grade | Baseline, 30 min
  Conjunctivocorneal epithelial staining will be assessed under a slit-lamp:
  Conjunctivocorneal epithelial staining will be assess corneal and conjunctival epithelium damage. Double vital staining approach with two microliters of a preservative-free solution containing 1% lissamine green and 1% sodium fluorescein will be instilled in the conjunctival sac.
  The eye will be sectioned into three equal pieces (temporal conjunctiva, cornea, and nasal conjunctiva). Each region receives a maximum staining score of three points and a minimum of zero points. The combined scores from all three parts were then recorded on a scale ranging from 0 (normal) to 9 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Eric Pazo, Study Chair — He Eye Hospital, Shenyang, China
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma J, Pazo EE, Zou Z, Jin F. Prevalence of symptomatic dry eye in breast cancer patients undergoing systemic adjuvant treatment: A cross-sectional study. Breast. 2020 Oct;53:164-171. doi: 10.1016/j.breast.2020.07.009. Epub 2020 Aug 5. PMID 32836200
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Heidari M, Noorizadeh F, Wu K, Inomata T, Mashaghi A. Dry Eye Disease: Emerging Approaches to Disease Analysis and Therapy. J Clin Med. 2019 Sep 11;8(9):1439. doi: 10.3390/jcm8091439. PMID 31514344
- [Background] Wang MTM, Feng J, Wong J, Turnbull PR, Craig JP. Randomised trial of the clinical utility of an eyelid massage device for the management of meibomian gland dysfunction. Cont Lens Anterior Eye. 2019 Dec;42(6):620-624. doi: 10.1016/j.clae.2019.07.008. Epub 2019 Jul 26. PMID 31358441
- [Background] Tichenor AA, Cox SM, Ziemanski JF, Ngo W, Karpecki PM, Nichols KK, Nichols JJ. Effect of the Bruder moist heat eye compress on contact lens discomfort in contact lens wearers: An open-label randomized clinical trial. Cont Lens Anterior Eye. 2019 Dec;42(6):625-632. doi: 10.1016/j.clae.2019.09.005. Epub 2019 Oct 3. PMID 31587960
- [Background] Olson MC, Korb DR, Greiner JV. Increase in tear film lipid layer thickness following treatment with warm compresses in patients with meibomian gland dysfunction. Eye Contact Lens. 2003 Apr;29(2):96-9. doi: 10.1097/01.ICL.0000060998.20142.8D. PMID 12695712
- [Background] Butovich IA. Lipidomics of human Meibomian gland secretions: Chemistry, biophysics, and physiological role of Meibomian lipids. Prog Lipid Res. 2011 Jul;50(3):278-301. doi: 10.1016/j.plipres.2011.03.003. Epub 2011 Mar 31. PMID 21458488
- [Background] McMonnies CW. Management of chronic habits of abnormal eye rubbing. Cont Lens Anterior Eye. 2008 Apr;31(2):95-102. doi: 10.1016/j.clae.2007.07.008. Epub 2008 Mar 19. PMID 18356094
- [Background] Zhang Q, Wu Y, Song Y, Qin G, Yang L, Talwar SS, Lin T, Talwar GDS, Zhang H, Xu L, Moore JE, Pazo EE, He W. Screening Evaporative Dry Eyes Severity Using an Infrared Image. J Ophthalmol. 2021 Aug 24;2021:8396503. doi: 10.1155/2021/8396503. eCollection 2021. PMID 34484814
- [Derived] Chen J, Yu S, Qin G, Moutari S, Moore JE, Xu L, He W, Pazo EE, He X. Immediate sequential changes in the tear film lipid layer following eyelid massage in dry eye syndrome: A comparative control study. Heliyon. 2024 Aug 20;10(17):e36590. doi: 10.1016/j.heliyon.2024.e36590. eCollection 2024 Sep 15. PMID 39286233